CLINICAL TRIAL: NCT02665793
Title: Mechanisms Underlying the Change in Threshold or Severity of Peanut-allergic Reactions in TRACE Peanut Study Participants - Extension Study
Brief Title: Mechanisms Underlying Peanut Allergic Reactions in TRACE Peanut Study Participants: Extension Study
Acronym: TRACEextension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Manchester (Other); Food Standards Agency, United Kingdom (Other Government); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Paul Turner, Clinician Scientist and Hon Consultant in Paediatric Allergy & Immunology, Imperial College London
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 15SM2445 vs4.1 27.12.2015; FP7-KBBE 312147 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Food Hypersensitivity; Peanut Hypersensitivity
Keywords: Peanut allergy; Food allergy; Thresholds; Anaphylaxis
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBPCFC to peanut cookie, then single-dose DBPCFC x 2 (Experimental): Patients will undergo 3 sets of double-blind, placebo-controlled food challenge (DBPCFC):
  1. DBPCFC to incremental doses of peanut (or placebo) baked into a cookie biscuit
  2. DBPCFC to a single dose of peanut (or placebo) equivalent to 1 dosing interval below that to which that patient reacted at the baseline DBPCFC to gain entry to the study, on two separate occasions
  Interventions: Other: DBPCFC to peanut cookie; Other: Single-dose DBPCFC to peanut flour; Other: Single-dose DBPCFC to peanut butter
- Single dose DBPCFC x 2, then DBPCFC to peanut cookie (Experimental): Patients will undergo 3 sets of double-blind, placebo-controlled food challenge (DBPCFC):
  1. DBPCFC to a single dose of peanut (or placebo) equivalent to 1 dosing interval below that to which that patient reacted at the baseline DBPCFC to gain entry to the study, on two separate occasions
  2. DBPCFC to incremental doses of peanut (or placebo) baked into a cookie biscuit
  Interventions: Other: DBPCFC to peanut cookie; Other: Single-dose DBPCFC to peanut flour; Other: Single-dose DBPCFC to peanut butter

INTERVENTIONS:
Other: DBPCFC to peanut cookie
Other: Single-dose DBPCFC to peanut flour — Single-dose DBPCFC to peanut in a water-continuous matrix, at a cumulative dose one dosing level below that individual's threshold (established at the baseline challenge). If no reaction is seen, participants will be given the next dosing level.
Other: Single-dose DBPCFC to peanut butter — Single-dose DBPCFC to peanut in a water-continuous matrix, at a cumulative dose one dosing level below that individual's threshold (established at the baseline challenge). If no reaction is seen, participants will be given the next dosing level.

SUMMARY:
Food allergy affects up to 10% of the population. The mainstay of management involves dietary avoidance and provision of rescue medication in the event of an accidental reaction. The Integrated approaches to food allergen and allergy management (iFAAM) collaboration is an EU-funded academic/clinical/industry consortium with the aim to improve allergen risk management including food labelling. Much of this work requires the validation of the minimum 'eliciting dose' for the food-allergic population and how this can be translated into risk management.

A number of studies (including iFAAM and the TRACE study - NCT01429896) have assessed the eliciting dose for peanut allergic patients, using food challenges where peanut-allergic individuals are eat incremental doses of peanut under strict medical supervision.

In this extension study, peanut-allergic subjects will have undergone (in a cross-over manner) three double-blind, placebo-controlled food challenges to peanut:

1. incremental doses of peanut in a water-continuous matrix;
2. incremental doses of peanut baked into a cookie biscuit;
3. a single dose of peanut in a water-continuous matrix.

The differences in eliciting dose, symptom pattern and underlying physiological mechanisms will provide essential data on how the presentation and consumption of peanut affects the amount needed to trigger an allergic reaction, to inform industry and food regulators as to how to best protect the food-allergic population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male and female participants in the TRACE study (NCT01429896) who are 18-45 years of age at the time of entry to the TRACE study (Visit 1) and had a positive DBPCFC to peanut at baseline (Visit 1).

Exclusion criteria

* unable to comply with study procedures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Minimum eliciting dose | 2 hours
  Minimum eliciting dose of peanut to trigger an objective allergic reaction according to international consensus criteria (PRACTALL))

SECONDARY OUTCOMES:
Symptom pattern | 12 hours
  Symptoms experienced following peanut challenge (defined according to international consensus criteria (PRACTALL) )

CONTACTS AND LOCATIONS:
Overall Officials: Clare Mills, PhD, Study Chair — University of Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made public through the Integrated approaches to food allergen and allergy management (iFAAM) collaboration

REFERENCES:
- [Derived] Turner PJ, Ruiz-Garcia M, Patel N, Abrantes G, Burrell S, Vazquez-Ortiz M, Skypala I, Durham SR, Boyle RJ. Delayed symptoms and orthostatic intolerance following peanut challenge. Clin Exp Allergy. 2021 May;51(5):696-702. doi: 10.1111/cea.13865. Epub 2021 Mar 21. PMID 33715235
- See also: iFAAM website — http://www.inflammation-repair.manchester.ac.uk/iFAAM/